CLINICAL TRIAL: NCT04558528
Title: Clinical Validation of Novel Malaria Diagnostic Tools for Point-of-Care Testing
Brief Title: Innovation Platform
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: MA014
Record Dates: First submitted 2020-09-15; First posted 2020-09-22 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Novel in vitro diagnostics and medical applications — Novel in vitro diagnostics and medical applications

SUMMARY:
In this study, a prospective evaluation of novel malaria diagnostic tools under development will be performed in malaria-endemic countries to assess their clinical performance for detection of malaria at point-of-care (POC). This study aims to support product development efforts and aims to provide early stage (TLR~5) technology developers with valuable information on performance and basic feasibility data that can help to accelerate development.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 years or older
* Presenting at the study site with symptoms and signs suggestive of malaria
* Freely agreeing to participate by signing an informed consent form (adults aged 18 and older and parent/legal guardian of a child) and providing assent (children aged 13-17)
* Willing to provide sample at enrolment

Exclusion Criteria:

* Presence of symptoms and signs of severe disease and/or central nervous system infections, as defined by WHO guidelines

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with symptoms suggestive of malaria seeking clinical care in health facilities
Sampling Method: Non-Probability Sample
Enrollment: 640 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Clinical performance assessment | up to 6 months
  Point estimates of clinical performance characteristics with 95% confidence intervals (sensitivity, specificity, NPV, PPV, and DOR) of nPOC using nPCR as reference for detecting malaria in patients with symptoms suggestive of malaria
Concordance | up to 6 months
  Point estimate with 95% confidence intervals of the percentage agreement in interpreting malaria diagnostics between the app and visual reading

CONTACTS AND LOCATIONS:
Locations (2):
- Eijkman Institute for Molecular Biology, Jakarta, Indonesia
- Stansile, Kigali, Rwanda